CLINICAL TRIAL: NCT04225884
Title: DTx for Pain: Behavioural Revalidation in Augmented and Virtual Reality for Chronic Pain; and Exploratory Pilot Study of a Virtual Reality Software
Brief Title: Digital Therapeutics (DTx) for Pain: Pilot Study of a Virtual Reality Software for Chronic Pain
Acronym: VIRPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 3129002
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DTx for pain (Active Comparator): Treatment A software
  Interventions: Other: DTx for pain software
- Control (Sham Comparator): Treatment B software
  Interventions: Other: Control software
- Standard care (Other): Pain medication
  Interventions: Other: Standard care

INTERVENTIONS:
Other: DTx for pain software — Software with active intervention
  Arms: DTx for pain
Other: Control software — Software without active intervention
  Arms: Control
Other: Standard care — Pain medication
  Arms: Standard care

SUMMARY:
Prospective, randomised, double-blind, 3-arm parallel group comparison of 2 different virtual reality softwares and standard care.

DETAILED DESCRIPTION:
Prospective, randomised, double-blind, 3-arm parallel group comparison of DTx for pain (treatment A), control (treatment B) and an open standard care arm, over 6-8 weeks. An optional adaptive, multi-objective, multi-purpose, extension is included. Study devices will be delivered to the patient's home with instructions for use; patients will receive remote technical support.

ELIGIBILITY:
Inclusion Criteria:

* Competent male or female adults (age ≥ 18 years).
* Chronic low back pain
* Written informed consent
* Finnish speaking
* having a clear, flat surface of at least 2 x 2 m of size to interact with DTx for pain
* Can stoop without severe pain

Exclusion Criteria:

* History of epilepsy, migraine, vertigo or psychosis
* Confirmed diagnosis of cancer
* Prone to strong motion sickness requiring treatment
* Pregnancy
* Physiotherapy based interventions contraindicated
* Severe or acute structural pathologies (e.g. spondylitis, epidural abscess, spondylolisthesis, acute herniated or ruptured disc, traumatic injury, or severe spinal stenosis) that could be worsened by the intervention as assessed by the principal investigator
* Has received (in last 2 years) or is receiving formal psychotherapy from a psychologist for pain or allied health care professional at the screening stage
* Any other condition that would affect posture or balance, and
* Prior participation in DTx for pain feasibility study or in any part of the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Self-report of disability, Oswestry | From randomisation upto 6-8 weeks
  Oswestry Disability Index (subjects with a score of ≤22 will be considered as responders), index 0%-100% (0=no disability, 100=maximum disability possible).
Self-report of disability; Pain Interference | From randomisation upto 6-8 weeks
  The Patient Reported Outcomes Information System (PROMIS) 6b - Pain Interference Scale, score 6-30 (6=pain not at all interfering patient's life, 30=maximum interfering to patient's life).
Objective report of disability, steps | From randomisation upto 6-8 weeks
  Average number of steps per day over one week, as assessed by wearable equipment, 0-maximum amount of steps (0=patient not taking steps at all, maximum disability; maximum number of steps=minimum disability).
Fear of movement and re-injury | From randomisation upto 6-8 weeks
  Tampa Scale of Kinesiophobia (TSK), score 17-68 (17=negligible or no kinesiophobia,68=extreme fear of pain with movement).
Pain Behaviour, pain intensity | From randomisation upto 6-8 weeks
  Numerical Rating Scale, PROMIS 3a - Pain Intensity Scale, score 3-15 (3=no pain,15=very severe pain).
Pain Behaviour, pain medications | From randomisation upto 6-8 weeks
  Any changes in pain medication during the study period are reported as outcome.
Quality of life, own experience | From randomisation upto 6-8 weeks
  EuroQol-5D-5L-scale: European Quality (EQ) of Life (l), 5-dimension-5-level-scale. a). Descriptive System, 5-dimension-5-level-scale, scores are converted to a value where 1 equals 'perfect health' and 0 equals 'dead'. b). Visual Analogue Score, score 0 to 100 where 100 is the best health you can imagine and 0 = the worst health you can imagine.
Quality of life, adverse events | From randomisation upto 6-8 weeks
  Adverse Event reporting, number of adverse events and their severity
Quality of life, change | From randomisation upto 6-8 weeks
  Patient Clinical Global Impression of Change (PGIC) results, score 1-7 (1=very much improved, 7=very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Orion Pharma Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- CPU Orion Pharma, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liikkanen S, Makinen M, Huttunen T, Sarapohja T, Stenfors C, Eccleston C. Body movement as a biomarker for use in chronic pain rehabilitation: An embedded analysis of an RCT of a virtual reality solution for adults with chronic pain. Front Pain Res (Lausanne). 2022 Dec 20;3:1085791. doi: 10.3389/fpain.2022.1085791. eCollection 2022. PMID 36606032
- [Derived] Eccleston C, Fisher E, Liikkanen S, Sarapohja T, Stenfors C, Jaaskelainen SK, Rice ASC, Mattila L, Blom T, Bratty JR. A prospective, double-blind, pilot, randomized, controlled trial of an "embodied" virtual reality intervention for adults with low back pain. Pain. 2022 Sep 1;163(9):1700-1715. doi: 10.1097/j.pain.0000000000002617. Epub 2022 Mar 25. PMID 35324507